CLINICAL TRIAL: NCT05523336
Title: Prospective Non-Interventional Trial to Evaluate Kinetics, Diagnostic and Prognostic Value of Pro-ADM as Compared to PCT in Patients Presenting With Infections or Other Complications Post Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Pro-ADM vs PCT in Patients With Complications Post Hematopoietic Stem Cell Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Prof, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: Trap-ADM
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stem Cell Transplant Complications
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample collection will be performed on T1 (first day of fever or day in ich a transplant-related complication is diagnosed), T2 (3 days after T1), T3 (10 days after T1). It will be analysed PCT and pro-ADM values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric patients receiving HCTS with infectious complications post HCTS: Paediatric patients receiving allogeneic hematopoietic stem cell transplantation (HCTS) and who present with infectious complications post HSCT or with transplant related complications (acute graft-versus-host disease- GvHD-, sinusoidal obstruction syndrome -SOS-, engraftment-ES- and pre-engraftment syndrome- pre-ES-, graft failure, thrombotic microangiopathy associated with HSCT- TA-TMA or those without complications post HSCT).
  Interventions: Other: observation
- Paediatric patients receiving HCTS without infectious complications post HCTS: Paediatric patients receiving HCTS without infectious complications post HCTS
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation and prospective data collection

SUMMARY:
Prospective, multicenter, spontaneous, non-interventional, non pharmacological. Study aimed at evaluate kinetics, diagnostic and prognostic value of pro-ADM (proadrenomedullin) as compared to PCT (procalcitonin) in patients presenting with infections or other complications post hematopoietic stem cell transplantation (HSCT)

DETAILED DESCRIPTION:
Evaluation of diagnostic performance of pro-ADM as compared to palliative care therapy (PCT) in paediatric and young adult patients with any type of complications after hematopoietic stem cell transplantation or with transplant related complications.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the parents/legal guardians and patient's assent/consent according to national regulations. For subjects who turn 18 years of age during participation in this study, participation in the future use portion of the study after their 18th birthday requires that they sign the informed consent statement following turning 18 years of age.
* Age at time of registration from 28 days to less than 39 years of age.
* Malignant disease (i.e. Acute lymphocytic leukemia (ALL), Acute myeloid leukemia (AML), Myelodysplastic syndromes (MDS)) or nonmalignant disease (e.g. immunodeficiency or inherited disorders of metabolism or hemoglobinopathies etc.) indicated for allogeneic HSCT.

Exclusion Criteria:

* Age less than 28 days
* Obese patients with body mass index: > 30 kg/m^2.
* Impaired cardiac function: severe cardiac insufficiency indicated by left ventricle ejection fraction (LVEF) ≤ 35%.
* Impaired liver function indicated by Bilirubin >3 times the upper limit of normal (ULN), or aspartate aminotransferase/alanine aminotransferase (AST/ALT) >10 times ULN
* Impaired renal function indicated by estimated glomerular filtration rate (GFR), according to the Schwartz formula for ages 1-17 and according to CDKEPI creatinine equation for ages above 17 years old) < 60 mL/min/1,73m^2.
* Concurrent severe active infection at the start of conditioning regimen

Ages: 28 Days to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and young adult patients affected by malignant or non-malignant disorders referred for HCST
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of diagnostic performance of pro-ADM as compared to PCT in patients receiving HSCT | 180 days after HSCT
  In order to achieve the objective, it will be considered paediatric and young adults patients affected by malignant/non-malignant disorders who have been subjected to HSCT and present with infectious complications post HSCT or with transplant related complications (acute graft-versus-host disease (GvHD), sinusoidal obstruction syndrome (SOS), engraftment (ES) and pre-engraftment syndrome (pre-E), graft failure, thrombotic microangiopathy associated with HSCT (TA-TMA) or those without complications post HSCT).

CONTACTS AND LOCATIONS:
Overall Officials: Franca Fagioli, MD, Principal Investigator — AOU Città della Salute e della Scienza di Torino - OIRM; Manuela Spadea, MD, Study Chair — AOU Città della Salute e della Scienza di Torino - OIRM
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin, Italy

IPD SHARING:
Plan to Share IPD: No